CLINICAL TRIAL: NCT03010527
Title: A Multicenter, 48-Week, Double-Blind, Placebo-Controlled, Parallel-Group Extension Study to Assess the Long-Term Safety, Tolerability, and Efficacy of Bimekizumab in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study to Evaluate the Long-term Safety, Tolerability and Efficacy of Bimekizumab in Patients With Chronic Plaque Psoriasis
Acronym: BE ABLE 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS0011; 2016-001892-57 (EudraCT Number)
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Results first posted 2021-10-25 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Chronic plaque psoriasis; Psoriasis; Bimekizumab
MeSH Terms: conditions — Psoriasis | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Subjects with a PASI90 response at Week 12 and receiving Placebo in PS0010 entering PS0011 will receive Placebo.
  Interventions: Other: Placebo
- Bimekizumab dosing regimen 1 (Experimental): Subjects with a PASI90 response at Week 12 receiving dosing regimen 1 in PS0010 entering PS0011 will receive the same dosing regimen.
  Subjects who do not achieve PASI90 response at Week 12 receiving dosing regimen 1 in PS0010 will be assigned to a higher dosing regimen.
  Interventions: Drug: Bimekizumab
- Bimekizumab dosing regimen 2 (Experimental): Subjects with a PASI90 response at Week 12 receiving dosing regimen 2 in PS0010 entering PS0011 will receive the same dosing regimen.
  Subjects who do not achieve PASI90 response at Week 12 receiving dosing regimen 2 in PS0010 will be assigned to a higher dosing regimen.
  Interventions: Drug: Bimekizumab
- Bimekizumab dosing regimen 3 (Experimental): Subjects that were initially randomized to bimekizumab dosage regimen 3, 4 and 5 in PS0010 will receive bimekizumab dosing regimen 3.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive bimekizumab injections every four weeks (Q4W)
  Other Names: UCB4940
  Arms: Bimekizumab dosing regimen 1; Bimekizumab dosing regimen 2; Bimekizumab dosing regimen 3
Other: Placebo — Subjects will receive Placebo injections every four weeks (Q4W)
  Arms: Placebo

SUMMARY:
This is a multicenter extension study to assess the long-term safety, tolerability and efficacy of bimekizumab in adult subjects with moderate to severe chronic plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent
* Subject completes all dosing requirements in feeder study and completes PS0010 study without meeting any withdrawal criteria
* Female subjects of childbearing potential and male subjects with a partner of childbearing potential must continue to use an acceptable method of contraception (as detailed in PS0010) for up to 20 weeks after the last dose of study treatment in PS0011

Exclusion Criteria:

* Subject has previously participated in this study.
* Female subjects who plan to become pregnant during the study or within 20 weeks following last dose of study medication. Male subjects who are planning a partner pregnancy during the study or within 20 weeks following the last dose
* Subject has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the subject's ability to participate in this study.
* Subject must have a negative interferon gamma release assay (IGRA) as measured at Week 8 of PS0010

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (36):
- United States (8):
  - Ps0011 708, Los Angeles, California
  - Ps0011 706, Washington D.C., District of Columbia
  - Ps0011 704, West Des Moines, Iowa
  - Ps0011 738, Wilmington, North Carolina
  - Ps0011 712, Portland, Oregon
  - Ps0011 733, Dallas, Texas
  - Ps0011 709, Houston, Texas
  - Ps0011 702, Houston, Texas
- Canada (6):
  - Ps0011 209, Edmonton
  - Ps0011 201, North Bay
  - Ps0011 206, Peterborough
  - Ps0011 214, Québec
  - Ps0011 203, Surrey
  - Ps0011 205, Waterloo
- Czechia (4):
  - Ps0011 300, Ostrava
  - Ps0011 303, Pardubice
  - Ps0011 301, Prague
  - Ps0011 304, Prague
- Hungary (3):
  - Ps0011 404, Kecskemét
  - Ps0011 400, Orosháza
  - Ps0011 405, Szekszárd
- Japan (4):
  - Ps0011 504, Chiyoda-ku
  - Ps0011 503, Minatoku
  - Ps0011 502, Nagoya
  - Ps0011 501, Shinagawa-ku
- Poland (11):
  - Ps0011 600, Bialystok
  - Ps0011 603, Bialystok
  - Ps0011 611, Bialystok
  - Ps0011 610, Gdynia
  - Ps0011 604, Kielce
  - Ps0011 608, Krakow
  - Ps0011 605, Lublin
  - Ps0011 606, Lublin
  - Ps0011 607, Warsaw
  - Ps0011 601, Wroclaw
  - Ps0011 609, Wroclaw

REFERENCES:
- [Result] Blauvelt A, Papp KA, Merola JF, Gottlieb AB, Cross N, Madden C, Wang M, Cioffi C, Griffiths CEM. Bimekizumab for patients with moderate to severe plaque psoriasis: 60-week results from BE ABLE 2, a randomized, double-blinded, placebo-controlled, phase 2b extension study. J Am Acad Dermatol. 2020 Nov;83(5):1367-1374. doi: 10.1016/j.jaad.2020.05.105. Epub 2020 May 29. PMID 32473974
- [Result] Gordon KB, Langley RG, Warren RB, Okubo Y, Stein Gold L, Merola JF, Peterson L, Wixted K, Cross N, Deherder D, Thaci D. Bimekizumab Safety in Patients With Moderate to Severe Plaque Psoriasis: Pooled Results From Phase 2 and Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2022 Jul 1;158(7):735-744. doi: 10.1001/jamadermatol.2022.1185. PMID 35544084
- See also: Product Information — https://www.ema.europa.eu/en/documents/product-information/bimzelx-epar-product-information_en.pdf
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in December 2016 and concluded in September 2018. Among the 217 participants in PS0011, no participants were assigned to receive placebo.
Pre-assignment Details: Participant Flow refers to the Full Analysis Set (FAS), which consisted of all enrolled participants who received at least 1 dose of the investigational medicinal product (IMP) and had a valid measurement of the primary efficacy variable at Baseline of PS0011.
Groups:
- Bimekizumab 64 mg Q4W: Participants received bimekizumab 64 milligrams (mg) injections, sc every four weeks (Q4W). Participants who achieved PASI90 response at Week 12 and received bimekizumab 64 mg Q4W in PS0010, were assigned to bimekizumab 64 mg Q4W in PS0011. Participants who did not achieve PASI90 response at Week 12 and received bimekizumab 64 mg Q4W in PS0010, were assigned to bimekizumab 160 mg Q4W in PS0011.
- Bimekizumab 160 mg Q4W: Participants received bimekizumab 160 mg injections, sc every four weeks (Q4W). Participants who achieved PASI90 response at Week 12 and received bimekizumab 160 mg Q4W or bimekizumab 160 mg with loading dose (w/LD) Q4W in PS0010, were assigned to bimekizumab 160 mg Q4W in PS0011. Participants who did not achieve PASI90 response at Week 12 and received bimekizumab 160 mg Q4W or bimekizumab 160 mg w/LD Q4W in PS0010, were assigned to bimekizumab 320 mg Q4W in PS0011.
- Bimekizumab 320 mg Q4W: Participants received bimekizumab 320 mg injections, sc every four weeks (Q4W). Participants receiving bimekizumab 320 mg Q4W and bimekizumab 480 mg Q4W, in PS0010 were assigned to receive bimekizumab 320 mg Q4W in PS0011, regardless of their PASI90 response at Week 12 in PS0010.
Period: Overall Study
Arm/Group | Bimekizumab 64 mg Q4W | Bimekizumab 160 mg Q4W | Bimekizumab 320 mg Q4W
Started | 15 | 111 | 91
Completed | 15 | 92 | 75
Not Completed | 0 | 19 | 16
Not completed — Death | 0 | 0 | 1
Not completed — Adverse Event | 0 | 4 | 2
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 4
Not completed — WITHDRAWAL CRITERIA #9 | 0 | 4 | 6
Not completed — WITHDRAWAL CRITERIA #12 | 0 | 4 | 2
Not completed — PDILI and WITHDRAWAL CRITERIA #9 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refer to the Safety Set (SS) which consisted of all participants who received at least 1 dose of the investigational medicinal product (IMP) in PS0011.
Arm/Group | Bimekizumab 64 mg Q4W | Bimekizumab 160 mg Q4W | Bimekizumab 320 mg Q4W | Total Title
Number analyzed (Participants) | 15 | 111 | 91 | 217
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 2 | 3
  Between 18 and 65 years | 14 | 105 | 77 | 196
  >=65 years | 1 | 5 | 12 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (14.7) | 44.5 (12.8) | 43.5 (14.7) | 44.1 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 40 | 31 | 77
  Male | 9 | 71 | 60 | 140
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian /Alaskan native | 0 | 1 | 1 | 2
  Asian | 1 | 11 | 6 | 18
  Black | 1 | 0 | 1 | 2
  White | 13 | 99 | 83 | 195

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Events (TEAEs) Adjusted by Duration of Subject Exposure to Treatment
Description: Treatment-emergent Adverse Events (TEAEs) were defined as those events which started on or after the date of first dose of PS0011 investigational medicinal product (IMP), or events in which severity worsened on or after the date of first dose of PS0011 study medication. The exposure adjusted incidence rate (EAIR) is defined as the number of subjects (n) with a specific AE adjusted for the exposure and was scaled to 100 subject-years: where the numerator is the total number of subjects experiencing the AE and the denominator is the total time at risk scaled to 100 subject-years; that is, the total summation of individual subject-years at risk up to the first occurrence of the AE for subjects with that AE, and the total subject-years at risk for those subjects not experiencing that AE, divided by 100.
Time Frame: From Baseline until Safety Follow-Up Visit (up to Week 64)
Population: The Safety Set (SS) consisted of all participants who received at least 1 dose of the study medication in PS0011.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Groups:
- Bimekizumab 64 mg Q4W (SS): Participants received bimekizumab 64 milligrams (mg) injections, sc every four weeks (Q4W). Participants who achieved PASI90 response at Week 12 and received bimekizumab 64 mg Q4W in PS0010, were assigned to bimekizumab 64 mg Q4W in PS0011. Participants who did not achieve PASI90 response at Week 12 and received bimekizumab 64 mg Q4W in PS0010, were assigned to bimekizumab 160 mg Q4W in PS0011. Participants who received at least one dose of the IMP formed the Safety Set (SS).
- Bimekizumab 160 mg Q4W (SS): Participants received bimekizumab 160 mg injections, sc every four weeks (Q4W). Participants who achieved PASI90 response at Week 12 and received bimekizumab 160 mg Q4W or bimekizumab 160 mg with loading dose (w/LD) Q4W in PS0010, were assigned to bimekizumab 160 mg Q4W in PS0011. Participants who did not achieve PASI90 response at Week 12 and received bimekizumab 160 mg Q4W or bimekizumab 160 mg w/LD Q4W in PS0010, were assigned to bimekizumab 320 mg Q4W in PS0011. Participants who received at least one dose of the IMP formed the SS.
- Bimekizumab 320 mg Q4W (SS): Participants received bimekizumab 320 mg injections, sc every four weeks (Q4W). Participants receiving bimekizumab 320 mg Q4W and bimekizumab 480 mg Q4W, in PS0010 were assigned to receive bimekizumab 320 mg Q4W in PS0011, regardless of their PASI90 response at Week 12 in PS0010. Participants who received at least one dose of the IMP formed the SS.
Arm/Group | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 320 mg Q4W (SS)
Number analyzed (Participants) | 15 | 111 | 91
no. of new events per 100 subject-years | 110.68 [53.08 to 203.55] | 225.26 [182.88 to 274.53] | 206.82 [162.95 to 258.86]

2. Secondary Outcome: Percentage of Participants With Psoriasis Area Severity Index (PASI90) Response Over Time
Description: The PASI90 response assessments are based on at least 90% improvement in the PASI score from Baseline. It averages the redness, thickness, and scaliness of the psoriatic lesions (on a 0-4 scale) and weights the resulting score by the area of skin involved. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity. PASI90 response is defined to be equal to 1 if the percentage improvement from Baseline in the PASI scores is 90% or greater and 0 if the percentage improvement from Baseline is less than 90%. This Outcome Measure presents results relative to PS0010 Baseline starting at PS0011 Baseline by PS0010 Week 12 response status.
Time Frame: From Baseline during the Treatment Period (up to Week 48)
Population: The Full Analysis Set (FAS) consisted of all enrolled participants who received at least 1 dose of the study medication in PS0011 and had a valid efficacy measurement for Psoriasis Area and Severity Index (PASI) at Baseline of PS0011.
Measure: Number; unit: percentage of participants
Groups:
- Bimekizumab 64 mg Q4W/Bimekizumab 64 mg Q4W/R (FAS): Participants who achieved PASI90 response at Week 12 and received bimekizumab 64 mg Q4W in PS0010, were assigned to bimekizumab 64 mg Q4W in PS0011. Participants formed the Full Analysis Set (FAS).
- Bimekizumab 160 mg Q4W/Bimekizumab 160 mg Q4W/R (FAS): Participants who achieved PASI90 response at Week 12 and received bimekizumab 160 mg Q4W or bimekizumab 160 mg with loading dose (w/LD) Q4W in PS0010, were assigned to bimekizumab 160 mg Q4W in PS0011. Participants formed the FAS.
- Bimekizumab 320 mg Q4W/Bimekizumab 320 mg Q4W/R (FAS): Participants who achieved PASI90 response at Week 12 and received bimekizumab 320 mg Q4W in PS0010, were assigned to bimekizumab 320 mg Q4W in PS0011. Participants formed the FAS.
- Bimekizumab 480 mg Q4W/Bimekizumab 320 mg Q4W/R (FAS): Participants who achieved PASI90 response at Week 12 and received bimekizumab 480 mg Q4W in PS0010, were assigned to bimekizumab 320 mg Q4W in PS0011. Participants formed the FAS.
- Placebo/Bimekizumab 160 mg Q4W/NR (FAS): Participants who did not achieve PASI90 response at Week 12 and received placebo Q4W in PS0010, were assigned to bimekizumab 160 mg Q4W in PS0011. Participants formed the FAS.
- Bimekizumab 64 mg Q4W/Bimekizumab 160 mg Q4W/NR (FAS): Participants who did not achieve PASI90 response at Week 12 and received bimekizumab 64 mg Q4W in PS0010, were assigned to bimekizumab 160 mg Q4W in PS0011. Participants formed the FAS.
- Bimekizumab 160 mg Q4W/Bimekizumab 320 mg Q4W/NR (FAS): Participants who did not achieve PASI90 response at Week 12 and received bimekizumab 160 mg Q4W or bimekizumab 160 mg w/LD Q4W in PS0010, were assigned to bimekizumab 320 mg Q4W in PS0011. Participants formed the FAS.
- Bimekizumab 320 mg Q4W/Bimekizumab 320 mg Q4W/NR (FAS): Participants who did not achieve PASI90 response at Week 12 and received bimekizumab 320 mg Q4W in PS0010, were assigned to bimekizumab 320 mg Q4W in PS0011. Participants formed the FAS.
- Bimekizumab 480 mg Q4W/Bimekizumab 320 mg Q4W/NR (FAS): Participants who did not achieve PASI90 response at Week 12 and received bimekizumab 480 mg Q4W in PS0010, were assigned to bimekizumab 320 mg Q4W in PS0011. Participants formed the FAS.
Arm/Group | Bimekizumab 64 mg Q4W/Bimekizumab 64 mg Q4W/R (FAS) | Bimekizumab 160 mg Q4W/Bimekizumab 160 mg Q4W/R (FAS) | Bimekizumab 320 mg Q4W/Bimekizumab 320 mg Q4W/R (FAS) | Bimekizumab 480 mg Q4W/Bimekizumab 320 mg Q4W/R (FAS) | Placebo/Bimekizumab 160 mg Q4W/NR (FAS) | Bimekizumab 64 mg Q4W/Bimekizumab 160 mg Q4W/NR (FAS) | Bimekizumab 160 mg Q4W/Bimekizumab 320 mg Q4W/NR (FAS) | Bimekizumab 320 mg Q4W/Bimekizumab 320 mg Q4W/NR (FAS) | Bimekizumab 480 mg Q4W/Bimekizumab 320 mg Q4W/NR (FAS)
Number analyzed (Participants) | 15 | 55 | 33 | 30 | 37 | 19 | 14 | 6 | 8
percentage of participants
  PS0011 Baseline | 100 | 100 | 100 | 100 | 0 | 0 | 0 | 0 | 0
  Week 4 | 100 | 100 | 97.0 | 100 | 45.9 | 42.1 | 42.9 | 66.7 | 50.0
  Week 8 | 100 | 96.4 | 100 | 100 | 67.6 | 73.7 | 57.1 | 83.3 | 50.0
  Week 12 | 100 | 96.4 | 100 | 96.7 | 81.1 | 78.9 | 64.3 | 100 | 62.5
  Week 16 | 100 | 92.7 | 100 | 96.7 | 83.8 | 78.9 | 64.3 | 100 | 62.5
  Week 20 | 100 | 89.1 | 93.9 | 96.7 | 89.2 | 84.2 | 78.6 | 83.3 | 62.5
  Week 24 | 100 | 85.5 | 97.0 | 96.7 | 83.8 | 78.9 | 71.4 | 83.3 | 75.0
  Week 28 | 93.3 | 90.9 | 97.0 | 96.7 | 91.9 | 84.2 | 71.4 | 83.3 | 50.0
  Week 32 | 100 | 89.1 | 97.0 | 93.3 | 91.9 | 73.7 | 71.4 | 83.3 | 50.0
  Week 36 | 100 | 85.5 | 97.0 | 93.3 | 91.9 | 73.7 | 71.4 | 66.7 | 50.0
  Week 40 | 100 | 83.6 | 87.9 | 86.7 | 89.2 | 78.9 | 71.4 | 83.3 | 50.0
  Week 44 | 100 | 81.8 | 87.9 | 86.7 | 89.2 | 78.9 | 71.4 | 83.3 | 50.0
  Week 48 | 100 | 80.0 | 87.9 | 86.7 | 91.9 | 68.4 | 71.4 | 66.7 | 50.0

3. Secondary Outcome: Percentage of Participants With Investigator´s Global Assessment Response (Clear or Almost Clear With at Least a 2 Category Improvement From Baseline on a 5-point Scale) Over Time
Description: The Investigator's Global Assessment (IGA) measures the overall severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild thickening, pink to light red coloration and predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4= severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA response is defined as clear (0) or almost clear (1) with at least a two category improvement from Baseline. This Outcome Measure presents results relative to PS0010 Baseline starting at PS0011 Baseline by PS0010 Week 12 response status.
Time Frame: From Baseline during the Treatment Period (up to Week 48)
Population: The FAS consisted of all enrolled participants who received at least 1 dose of the study medication in PS0011 and had a valid efficacy measurement for PASI at Baseline of PS0011.
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 64 mg Q4W/Bimekizumab 64 mg Q4W/R (FAS) | Bimekizumab 160 mg Q4W/Bimekizumab 160 mg Q4W/R (FAS) | Bimekizumab 320 mg Q4W/Bimekizumab 320 mg Q4W/R (FAS) | Bimekizumab 480 mg Q4W/Bimekizumab 320 mg Q4W/R (FAS) | Placebo/Bimekizumab 160 mg Q4W/NR (FAS) | Bimekizumab 64 mg Q4W/Bimekizumab 160 mg Q4W/NR (FAS) | Bimekizumab 160 mg Q4W/Bimekizumab 320 mg Q4W/NR (FAS) | Bimekizumab 320 mg Q4W/Bimekizumab 320 mg Q4W/NR (FAS) | Bimekizumab 480 mg Q4W/Bimekizumab 320 mg Q4W/NR (FAS)
Number analyzed (Participants) | 15 | 55 | 33 | 30 | 37 | 19 | 14 | 6 | 8
percentage of participants
  PS0011 Baseline | 100 | 96.4 | 100 | 100 | 5.4 | 10.5 | 35.7 | 50.0 | 25.0
  Week 4 | 100 | 98.2 | 97.0 | 100 | 56.8 | 57.9 | 42.9 | 66.7 | 62.5
  Week 8 | 100 | 96.4 | 97.0 | 100 | 75.7 | 84.2 | 57.1 | 83.3 | 62.5
  Week 12 | 100 | 92.7 | 97.0 | 96.7 | 81.1 | 89.5 | 64.3 | 83.3 | 62.5
  Week 16 | 100 | 90.9 | 97.0 | 96.7 | 83.8 | 78.9 | 57.1 | 66.7 | 62.5
  Week 20 | 100 | 85.5 | 93.9 | 96.7 | 89.2 | 84.2 | 71.4 | 66.7 | 75.0
  Week 24 | 100 | 81.8 | 97.0 | 93.3 | 83.8 | 84.2 | 64.3 | 83.3 | 62.5
  Week 28 | 93.3 | 89.1 | 97.0 | 93.3 | 86.5 | 84.2 | 71.4 | 66.7 | 62.5
  Week 32 | 100 | 85.5 | 93.9 | 93.3 | 89.2 | 78.9 | 71.4 | 66.7 | 50.0
  Week 36 | 100 | 81.8 | 90.9 | 93.3 | 86.5 | 78.9 | 71.4 | 66.7 | 37.5
  Week 40 | 100 | 83.6 | 87.9 | 86.7 | 86.5 | 78.9 | 71.4 | 66.7 | 50.0
  Week 44 | 100 | 81.8 | 87.9 | 86.7 | 83.8 | 78.9 | 71.4 | 66.7 | 50.0
  Week 48 | 100 | 78.2 | 87.9 | 86.7 | 89.2 | 68.4 | 71.4 | 66.7 | 62.5

ADVERSE EVENTS:
Time Frame: From PS0011 Baseline and up to Safety-Follow Up (SFU) (up to Week 64)
Arm/Group | Bimekizumab 64 mg Q4W (SS) | Bimekizumab 160 mg Q4W (SS) | Bimekizumab 320 mg Q4W (SS)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/111 | 2/91
Serious Adverse Events (participants affected / at risk) | 1/15 | 7/111 | 7/91
Other Adverse Events (participants affected / at risk) | 10/15 | 56/111 | 51/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimekizumab 64 mg Q4W (SS) (N=15) | Bimekizumab 160 mg Q4W (SS) (N=111) | Bimekizumab 320 mg Q4W (SS) (N=91)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Otitis externa bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
IgA nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Uterine cervix stenosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimekizumab 64 mg Q4W (SS) (N=15) | Bimekizumab 160 mg Q4W (SS) (N=111) | Bimekizumab 320 mg Q4W (SS) (N=91)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (2) | 13 (17) | 15 (19)
Skin candida (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Angular cheilitis (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (4) | 15 (20) | 11 (14)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 10 (12) | 9 (12)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (1) | 1 (2)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Gamma-glutamyl-transferase increased (Investigations) | 1 (1) | 4 (6) | 3 (4)
Hyperphagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 6 (7)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6) | 6 (8)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (6) | 3 (3)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 2 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6) | 5 (5)
Hypertension (Vascular disorders) | 2 (2) | 8 (10) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT03010527/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT03010527/SAP_001.pdf